CLINICAL TRIAL: NCT04629131
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Following Intramuscular Administration of a Single Dose of TNM002 in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TNM002 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhuhai Trinomab Pharmaceutical Co., Ltd. (Industry)
Collaborators: TIGERMED AUSTRALIA PTY LIMITED (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TNM002-P1-AU01
Record Dates: First submitted 2020-11-05; First posted 2020-11-16 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Healthy Adult Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 TNM002 10 μg/kg/Placebo (Experimental): Sentinel dosing will be conducted for Cohort 1. Two participants will be dosed (1 with TNM002, 1 with placebo) at least 72 hours prior to subsequent dosing. The remaining participants will only be dosed if no significant safety signals are identified in the sentinel participants. In total, eight subjects will be randomly assigned to receive either TNM002 or placebo at a 3:1 ratio (i.e. 6 subjects receive TNM002 and 2 with placebo).
  Interventions: Biological: TNM002 Dosage 1 (10 μg/kg); Biological: Placebo
- Cohort 2 TNM002 35 μg/kg/Placebo (Experimental): Eight subjects will be randomly assigned to receive either TNM002 or placebo at a 3:1 ratio (i.e. 6 subjects receive TNM002 and 2 with placebo).
  Interventions: Biological: TNM002 Dosage 2 (35 μg/kg); Biological: Placebo
- Cohort 3 TNM002 100 μg/kg/Placebo (Experimental): Eight subjects will be randomly assigned to receive either TNM002 or placebo at a 3:1 ratio (i.e. 6 subjects receive TNM002 and 2 with placebo).
  Interventions: Biological: TNM002 Dosage 3 (100 μg/kg); Biological: Placebo
- Cohort 4 TNM002 250 μg/kg/Placebo (Experimental): Eight subjects will be randomly assigned to receive either TNM002 or placebo at a 3:1 ratio (i.e. 6 subjects receive TNM002 and 2 with placebo).
  Interventions: Biological: TNM002 Dosage 4 (250 μg/kg); Biological: Placebo

INTERVENTIONS:
Biological: TNM002 Dosage 1 (10 μg/kg) — TNM002 (human monoclonal antibody against tetanus toxin), 10 μg/kg, Intramuscular injection, given once.
  Arms: Cohort 1 TNM002 10 μg/kg/Placebo
Biological: Placebo — placebo to match TNM002 Dosage 1, given once
  Arms: Cohort 1 TNM002 10 μg/kg/Placebo
Biological: TNM002 Dosage 2 (35 μg/kg) — TNM002 (human monoclonal antibody against tetanus toxin), 35 μg/kg, Intramuscular injection, given once
  Arms: Cohort 2 TNM002 35 μg/kg/Placebo
Biological: Placebo — placebo to match TNM002 Dosage 2, given once
  Arms: Cohort 2 TNM002 35 μg/kg/Placebo
Biological: TNM002 Dosage 3 (100 μg/kg) — TNM002 (human monoclonal antibody against tetanus toxin), 100 μg/kg, Intramuscular injection, given once
  Arms: Cohort 3 TNM002 100 μg/kg/Placebo
Biological: Placebo — placebo to match TNM002 Dosage 3, given once
  Arms: Cohort 3 TNM002 100 μg/kg/Placebo
Biological: TNM002 Dosage 4 (250 μg/kg) — TNM002 (human monoclonal antibody against tetanus toxin), 250 μg/kg, Intramuscular injection, given once
  Arms: Cohort 4 TNM002 250 μg/kg/Placebo
Biological: Placebo — placebo to match TNM002 Dosage 4, given once
  Arms: Cohort 4 TNM002 250 μg/kg/Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics properties of TNM002 following a single intramuscular dose in healthy adult subjects.

DETAILED DESCRIPTION:
The study a randomized, double-blinded, placebo-controlled, dose-escalation phase I trial. A total of 32 healthy adult subjects will be enrolled into 4 cohorts sequentially. Each participant will receive a single IM dose of TNM002 or placebo according to the cohort in which they were enrolled. After injection (Day 1), participants remain in the study site for observation up to 5 days. Following completion of the safety assessments and sampling for PK/PD analyses on Day 4, participants will be discharged from the study site. On Day 8, 15, 29, 43, 64 and 85, participants will return for safety assessments.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet the following criteria to be enrolled in this study:

1. Healthy male or female, 18-55 years of age (both inclusive);
2. Able to give signed written informed consent form;
3. Able to well communicate with investigators as well as understand and adhere to the requirements of this study.
4. Body mass index (BMI, weight [kg]/height [m]2) within 18.0-32.0 kg/m2 (both inclusive);
5. Blood Pressure (BP) and 12-lead ECG showing no clinically significant abnormalities at the discretion of the Principal Investigator during screening;
6. Subjects having no clinically significant abnormality on physical examination, clinical laboratory tests, liver function or kidney function as determined by Principal Investigator (PI);
7. Females must be either under surgical sterile (i.e. had a bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 6 months before the first dose of study drug) or under postmenopausal for at least 1 year before the first dose of study drug or agree to use an acceptable method of contraception from screening until 90 days after last study drug administration. Males who are sexually active and who are partners of women of childbearing potential must agree to use effective contraception from screening until 90 days after last drug administration.

   * acceptable method of contraception

     * Use of intrauterine device
     * Use of oral, injected or implanted hormonal methods of contraception
     * Concomitant use of barrier contraception method
     * Surgical contraception methods (e.g., vasectomy, salpingectomy, hysterectomy, etc.)

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. History or evidence of severe drug or excipient allergy, or hypersensitivity to other therapeutic mAbs;
2. History or evidence of autoimmune disease or possible immunodeficiency state, including positive screening test for HIV;
3. History or evidence of chronic hepatitis, including positive screening test for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody;
4. History or evidence of tetanus infection, or exposure to tetanus vaccine within 6 months prior to the fist drug administration;
5. Exposure to any live attenuated vaccine within 4 weeks prior to the fist drug administration;
6. Exposure to any inactivated vaccine within 2 weeks prior to the fist drug administration;
7. History or evidence of any other acute or chronic disease that, in the opinion of the investigator, may have interfered with the evaluation of the safety or immunogenicity of the drug or compromised the safety of the subject; for example, a clinically relevant history of respiratory, thyroid, gastrointestinal, renal, hepatic, hematological, lymphatic, oncologic, cardiovascular, psychiatric, neurological, musculoskeletal, genitourinary, infective, inflammatory, immunological, dermatological, or connective tissue disease
8. Subjects with surgery (except for minor outpatient surgery) within past 3 months prior to screening, or planned surgery during study;
9. Subjects with intolerance or insufficient venous access to permit regular venepuncture;
10. Known or suspected history of drug abuse within the past 5 years or with positive urine drug test at the screening;
11. Donated blood >400 mL or significant blood loss equivalent to 400 mL or received blood transfusion within 3months of screening; or donated blood >200 mL or significant blood loss equivalent to 200 mL within 1 month prior to the screening;
12. Participation in any other clinical studies with chemical or biological drugs or device within 4 weeks or 5 times the half-life of the specific drug/biologics (whichever is longer), prior to the first drug administration;
13. Use of any other drug, including over-the-counter medications, herb medicines within 14 days prior to the first drug administration (except for contraceptive medication in WOCBP, or concomitant medications that are considered necessary for the subject's welfare and unlikely to interfere with the study);
14. Receipt of an Ig or blood product within 90 days prior to the first drug administration;
15. Receipt of immunosuppressive medications, other than inhaled or topical immunosuppressant drugs, within 45 days prior to the first drug administration;
16. Habitual use of nicotine products or smoking within 3 months (more than 5 cigarettes per day) prior to screening or unwilling to refrain from nicotine products during study participation;
17. History of significant alcohol abuse within 6 months of screening or any indication of regular use of more than 14 units of alcohol per week (1 Unit=360 mL of beer or 45 mL of alcohol 40% or 150 mL of wine) or taking a product containing alcohol 2 days prior to dosing, or having a positive alcohol breath test during the screen period.;
18. Malignancy within 5 years of screening visit (except basal cell skin carcinoma);
19. Subject who is considered unsuitable for participating in the study in the opinion of investigator;
20. Nursing mothers or pregnant women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Up to 105 days post dosing
  The investigator will assess the intensity for each AE reported during the study based on the investigator's clinical judgment. Adverse events will be recorded according to CTCAE V5.0.
Clinically significant abnormality in physical examinations | Up to 105 days post dosing
  clinically significant abnormality in general condition, skin, eyes/ears/nose/mouth/throat, neck/thyroid, chest/lungs, heart, vascular system, lymph nodes, abdomen, extremities, nervous systems/reflexes, musculoskeletal, spine
Change in RR intervals (msec) | Up to 105 days post dosing
  Measured using a 12 Lead Electrocardiogram
Change in PR intervals (msec) | Up to 105 days post dosing
  Measured using a 12 Lead Electrocardiogram
Change in QRS duration (msec) | Up to 105 days post dosing
  Measured using a 12 Lead Electrocardiogram
Change in QT intervals (msec) | Up to 105 days post dosing
  Calculated using measurements by a 12 Lead Electrocardiogram
Change in QTcB intervals (msec) | Up to 105 days post dosing
  Calculated using measurements by a 12 Lead Electrocardiogram
Change in QTcF intervals (msec) | Up to 105 days post dosing
  Calculated using measurements by a 12 Lead Electrocardiogram
Change in Semi recumbent blood pressure (mmHg) | Up to 105 days post dosing
Change in pulse rate (bpm) | Up to 105 days post dosing
Change in body temperature (celsius) | Up to 105 days post dosing
Change in Hematocrit (ratio) | Up to 105 days post dosing
  Measured by hematology test
Change in Haemoglobin (g/L) | Up to 105 days post dosing
  Measured by hematology test
Change in Mean corpuscular hemoglobin (pg) | Up to 105 days post dosing
  Measured by hematology test
Change in Mean corpuscular hemoglobin concentration (g/L) | Up to 105 days post dosing
  Measured by hematology test
Change in Mean corpuscular volume (fL) | Up to 105 days post dosing
  Measured by hematology test
Change in Platelet count (cells x 10^9/L)) | Up to 105 days post dosing
  Measured by hematology test
Change in Red blood cell count (cells x 10^12/L) | Up to 105 days post dosing
  Measured by hematology test
Change in White blood cell count (cells x 10^9/L) | Up to 105 days post dosing
  Measured by hematology test
Change in differential leukocyte count (cells x 10^9/L) | Up to 105 days post dosing
  Including eosinophils, monocytes, lymphocytes, basophils, and neutrophils, Measured by hematology test
Change in Serum Alanine Aminotransferase (ALT) (U/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Serum Albumin (g/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Serum Alkaline Phosphatase (ALP) (U/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Serum Aspartate Aminotransferase (AST) (U/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Serum Total Bilirubin (umol/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Serum Blood urea nitrogen (BUN) (mmol/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Serum Calcium (mmol/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Serum Chloride (mmol/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Serum Cholesterol (mmol/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Serum Creatinine (umol/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Serum Creatine Kinase (U/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Serum Glucose (mmol/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Serum Lactate Dehydrogenase (U/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Serum Phosphorus (mmol/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Serum Potassium (mmol/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Serum Total protein (g/L) | Up to 105 days post dosing
  measured by serum chemistry
Change in Urine Bilirubin (U-BIL) | Up to 105 days post dosing
  measured by Urinalysis
Change in Urine Glucose (GLU) (mg/dL) | Up to 105 days post dosing
  measured by Urinalysis
Change in Urine erythrocytes (U-RBC) | Up to 105 days post dosing
  measured by Urinalysis
Change in Urinary leukocyte (U-LEU) | Up to 105 days post dosing
  measured by Urinalysis
Change in Urine nitrites (U-NIT) | Up to 105 days post dosing
  measured by Urinalysis
Change in Urine protein (U-PRO) | Up to 105 days post dosing
  measured by Urinalysis
Change in Urine specific gravity (U-SG) | Up to 105 days post dosing
  measured by Urinalysis
Change in Urine urobilinogen (URO) | Up to 105 days post dosing
  measured by Urinalysis
Change in Prothrombin time (sec) | Up to 105 days post dosing
  measured by Blood Coagulation test
Change in Activated partial thromboplastin time (APTT)(sec) | Up to 105 days post dosing
  measured by Blood Coagulation test
Change in fibrinogen (g/L) | Up to 105 days post dosing
  measured by Blood Coagulation test
Change in international normalized ratio (INR) | Up to 105 days post dosing
  measured by Blood Coagulation test

SECONDARY OUTCOMES:
Anti-TNM002 antibodies | Up to 105 days post dosing
  The numbers of subjects who developed anti-TNM002 antibodies
Anti-TNM002 antibodies | Up to 105 days post dosing
  The percentages of subjects who developed anti-TNM002 antibodies
Maximum observed plasma concentration (Cmax) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above
Time of maximum plasma concentration (Tmax) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above
Terminal half-life (T1/2) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above
Area under the plasma concentration-time curve from time-zero to the time of the last measurable concentration (AUC0-last) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above
Area under the plasma concentration-time curve from time-zero extrapolated to infinite time (AUC0-inf) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above
Apparent oral clearance (CL/F) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above
Apparent volume of distribution (Vz/F) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above
Mean retention time (MRT) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above
Lambda z - the reciprocal of elimination rate constant | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above
The ratio of area under the plasma concentration-time curve from time-zero to the time of the last measurable concentration (AUC0-last) extrapolated to AUC0-inf over AUC0-inf (% AUCex) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above

OTHER OUTCOMES:
Tetanus-antibody titer in serum | Up to 105 days post dosing
Time to achieve the maximum tetanus-antibody titer | Up to 105 days post dosing
The percentage of subjects with a change of titer ≥ 0.2 IU/mL from the baseline | Up to 105 days post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Lemech, FRACP, Principal Investigator — Scientia Clinical Research Ltd
Locations (1):
- Scientia Clinical Research, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in these articles, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Academics who provide a methodologically sound proposal.